CLINICAL TRIAL: NCT05758272
Title: Evaluation of a Workplace Smoking Cessation Program in Hong Kong: a Pragmatic Cluster Randomized Controlled Trial of Mobile Supported Simple Physical Exercise for Smoking Cessation
Brief Title: Evaluation of a Workplace Smoking Cessation Program in Hong Kong (Phase VI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCPW Phase 6
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Smokers; Workplace; Exercise
Keywords: smokers; Workplace; Exercise; mhealth; intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile phone-based simple physical exercise intervention (Experimental): Regular messages supporting participants in practicing simple physical exercises and assist in managing cravings will be sent to participants via IM apps and scheduled in a tapering manner for 3 months (twice per week in the first month to once per week in the third month). Images and videos explaining and demonstrating the simple physical exercises will be sent to the participants via IM apps, which serves as a reminder and supporting materials for participants. The benefits of exercise in SC will be explained. The investigators will also encourage the practice of moderate/ vigorous exercises to further improve the physical activity and well-being of the participants. Various delivery formats of messages will be considered to attract participants' interest such as text, emojis, voice, image, animation, and video. The simple exercises consist of a) Zero-time exercises (ZTEx), b) handgrip exercises and c) resistance exercises.
  Interventions: Behavioral: mobile phone-based simple physical exercise reminder to help quit smoking
- regular text-based intervention (Placebo Comparator): The control group will receive 6 regular messages via IM at twice per month within 3 months. These messages cover simple cessation advice and reminders for telephone follow-ups.
  Interventions: Behavioral: regular text-based intervention

INTERVENTIONS:
Behavioral: mobile phone-based simple physical exercise reminder to help quit smoking — Regular messages supporting participants in practicing simple physical exercises and assist in managing cravings will be sent to participants via IM apps and scheduled in a tapering manner for 3 months (twice per week in the first month to once per week in the third month). Images and videos explaining and demonstrating the simple physical exercises will be sent to the participants via IM apps, which serves as a reminder and supporting materials for participants. The benefits of exercise in SC will be explained. The investigator will also encourage the practice of moderate/ vigorous exercises to further improve the physical activity and well-being of the participants. Various delivery formats of messages will be considered to attract participants' interest such as text, emojis, voice, image, animation, and video. The simple exercises consist of a) Zero-time exercises (ZTEx), b) handgrip exercises and c) resistance exercises.
  Arms: mobile phone-based simple physical exercise intervention
Behavioral: regular text-based intervention — The control group will receive 6 regular messages via IM at twice per month within 3 months. These messages cover simple cessation advice and reminders for telephone follow-ups.
  Arms: regular text-based intervention

SUMMARY:
This study aims to test, by a 2-arm RCT, the effectiveness of an intervention that includes mobile phone-supported simple physical exercise for smoking cessation in workplaces in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18 or above
2. Smoke at least 1 cigarette per day or use other tobacco products (EC, HTP and others) daily
3. Able to communicate in Cantonese/Mandarin and read Chinese
4. Able to use instant messaging tools (e.g. WhatsApp) for communication
5. Stay in Hong Kong during the intervention and follow-up periods (12 months)

Exclusion Criteria:

1. Smokers who are psychologically or physically unable to communicate
2. Currently joining other smoking cessation program(s)
3. Smokers who cannot tolerate the proposed exercise program
4. Smokers who have severe mental illnesses

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 646 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported 7-day point-prevalence abstinence (PPA) at 6-months follow-up | at 6-month after treatment initiation (3 months after the end of treatment)
  Self-reported abstinence in the past 7 days at 6-months after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping WANG, PhD, Principal Investigator — School of Nursing, The University of Hong Kong Hong Kong, Hong Kong China
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Participant data (IPD) will only be used for data analysis by the investigators, kept strictly confidential, and not disclosed to anyone outside the research group.